CLINICAL TRIAL: NCT04307615
Title: Evaluation of Continous Positive Airway Pressure (CPAP) in Swimming Induced Pulmonary Edema (SIPE) -a Randomized Single-blinded Controlled Study
Brief Title: O2 Versus CPAP Treatment of Patients Undergoing SIPE Therapy (OCTOPUS)
Acronym: OCTOPUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Maria Hårdstedt, Dr. Maria Hårdstedt, PhD, Specialist Internal Medicine, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCTOPUS001
Record Dates: First submitted 2020-02-04; First posted 2020-03-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Swimming Induced Pulmonary Edema (SIPE); Pulmonary Edema; Lung Diseases
Keywords: continuous positive airway pressure (CPAP); oxygen; therapeutics; ultrasonography; oximetry
MeSH Terms: conditions — Pulmonary Edema; Lung Diseases | interventions — Oxygen; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen + CPAP-treatment (Experimental)
  Interventions: Combination Product: Oxygen + continuous positive airway pressure (CPAP)
- Oxygen-treatment (Active Comparator)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Combination Product: Oxygen + continuous positive airway pressure (CPAP) — Oxygen-driven CPAP (7,5 cmH2O): 20 min treatment followed by 10 min rest and assessment
  Arms: Oxygen + CPAP-treatment
Drug: Oxygen — Oxygen: 20 min treatment followed by 10 min rest and assessment
  Arms: Oxygen-treatment

SUMMARY:
In swimming induced pulmonary edema (SIPE), there is a lack of knowledge regarding optimal treatment. The present study was designed to assess the benefit of continuous positive airway pressure (CPAP) compared to oxygen as a first line treatment of SIPE in the out-of-hospital environment.

DETAILED DESCRIPTION:
Swimming induced pulmonary edema (SIPE) is an unusual condition affecting otherwise healthy swimmers. SIPE is characterized by acute onset of dyspnea and cough, excessive sputum and occasionally hemoptysis when swimming in open water. The condition usually resolves spontaneously within 48 hours, but may result in serious illness and require emergency care. Case reports describe acute treatment with oxygen alone or in combination with diuretics, beta-agonist-inhalation or continuous positive airway pressure (CPAP). Evidence for optimal treatment strategy is lacking. This study intends to determine whether oxygen alone or applied together with CPAP leads to improvement of oxygen saturation and recovery of patients. The aim is to treat patients on site without involving hospital care. We study a large cohort of approximately 12 000 swimmers during Vansbrosimningen, Sweden's biggest annual open water event with a yearly incidence of SIPE about 0,4%.

Adult patients clinically diagnosed with SIPE are randomly assigned in 2 groups receiving treatment during 20 minutes: (1) oxygen 10l/min or (2) oxygen 10l/min and CPAP 7,5 cm H2O. Assessment with outcome measures is taken 10 minutes after treatment. Primary endpoint: oxygen saturation (%) by pulse oxymetry.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of swimming induced pulmonary edema (SIPE) with need of acute treatment (oxygen saturation ≤91%)
* 18 years and older
* informed consent

Exclusion Criteria:

* declined consent
* suspected acute coronary syndrome
* severe asthma diagnosed together with pulmonary edema where beta-agonist-inhalation is needed prior to treatment of pulmonary edema
* hemodynamic instability or decreased consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Absolute peripheral oxygen saturation (%) after treatment | after 20 min treatment followed by 10 min rest
  Peripheral oxygen saturation % (continuous variable) measured by peripheral pulse oximetry

SECONDARY OUTCOMES:
Change in absolute peripheral oxygen saturation (%) before and after treatment | change before versus after 20 min treatment followed by 10 min rest
  Change in peripheral oxygen saturation % (continuous variable) measured by pulse oximetry before and after treatment
Recovery (yes/no) after treatment | after 20 min treatment followed by 10 min rest
  Recovery, defined by "peripheral oxygen saturation >95% after treatment" or no recovery, defined by "peripheral oxygen saturation ≤95% after treatment"
Interstitial syndrome assessed by lung ultrasound (yes/no) after treatment | after 20 min treatment followed by 10 min rest
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Bilateral or unilateral presence of two or more positive regions define positive interstitial syndrome.
Absolute number of regions presenting B-lines on lung ultrasound after treatment | after 20 min treatment followed by 10 min rest
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Assessment of the total number of positive regions.
Change in absolute number of regions presenting B-lines on lung ultrasound before and after treatment | change before versus after 20 min treatment followed by 10 min rest
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Assessment of the total number of positive regions. Change in absolute number of regions presenting B-lines on lung ultrasound before and after treatment
Change in patient reported outcome measures before and after treatment | change before versus after 20 min treatment followed by 10 min rest
  Six different patient reported outcome measures assessed by numeric rating scale (NRS) 0-10: cough, sputum, air hunger, breathing effort, tightness in chest, anxiousness. The patients will assess symptoms prior to and after treatment.
Admission to hospital (yes/no) | 2 hours
  admission to hospital within or after a maximal treatment time of 40 minutes followed by 20 min rest.
total treatment time | 2 hours
  total treatment time until oxygen saturation ≥96% is reached.
subgroup analysis | 1 hour
  treatment outcome analysis in patients with different baseline oxygen saturation on admission

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Clinical Research Dalarna, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No